CLINICAL TRIAL: NCT03843580
Title: Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) Could Decrease the Incidence of Oxygen Desaturation During Suspension Laryngoscopy: a Randomized Controlled Trial
Brief Title: Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) Could Decrease the Incidence of Oxygen Desaturation During Suspension Laryngoscopy: a Randomized Controlled Trial (Optilaryngo)
Acronym: optilaryngo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A00112-55
Record Dates: First submitted 2019-02-13; First posted 2019-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2020-02

CONDITIONS: Apnea, Postanesthetic; Desaturation of Blood; Apnea; Anesthesia; Larynx Disease; Pharynx; Anomaly
Keywords: Time of apnea; Optiflow; Thrive; Apnea oxygenation; Suspension laryngoscopy; General Anesthesia; Oxygenation apnea
MeSH Terms: conditions — Butyrylcholinesterase deficiency; Apnea; Laryngeal Diseases; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Allocation (No Intervention): apnea without oxygenation like usual traitement
- oxygenation optiflow (Experimental): optiflow oxygenation during apnea
  Interventions: Device: optiflow

INTERVENTIONS:
Device: optiflow — we use Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (thrive-optiflow) during general anesthesia for suspension laryngoscopy
  Arms: oxygenation optiflow

SUMMARY:
Suspension laryngoscopy is realised during apnea. In effect, surgeons are in the mouth of the patient and we can't have access at the aiways.

So investigators like to use a Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE) to increase time of apnea and decrease the impact of oxygen desaturation.

ELIGIBILITY:
Inclusion Criteria:

* suspension laryngoscopy

Exclusion Criteria:

* THRIVE contraindication:
* epistaxis
* undrained pneumothorax
* Recent gastroesophageal surgery (1months)
* Skull Fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
desaturation defined as the number of patient who presented at least one desaturation during suspension laryngoscopy | Two hours
  the number of patient who presented at least one desaturation during suspension laryngoscopy. An oxygen desaturation define like SpO2<96%

SECONDARY OUTCOMES:
hypoxemia (decrease the number of Hypoxemia event define like SpO2<90%) | 2 hours
  Decrease the number of Hypoxemia event define like SpO2<90%
side effect | 2 hours
  decrease the number of side effects

OTHER OUTCOMES:
time of apnea | 2 hours
  increase time of apnea with THRIVE

CONTACTS AND LOCATIONS:
Overall Officials: Eleonore Mulac-Vauclair, Principal Investigator — Centre Francois Baclesse; Pierre-Emmanuel Marsan, Principal Investigator — University Hospital, Caen; Kamga Herve, Principal Investigator — University Hospital, Caen; Boutros Mariam, Principal Investigator — University Hospital, Caen
Locations (2):
- France (2):
  - CaenUH, Caen, Normandy
  - Centre François Baclesse, Caen